CLINICAL TRIAL: NCT04631354
Title: A Phase One Open Label, Crossover Study in Healthy Adult Subjects to Quantify Lung Deposition and Distribution of 99mTc Radiolabelled S-770108 Inhalation Powder Formulation Delivered by a Novel Inhaler Device
Brief Title: Study in Healthy Adults to Quantify Lung Deposition and Distribution of Radio-labelled S-770108 Inhalation Powder Formulation Delivered by a Novel Inhaler Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1604P2111; 2018-004469-15 (EudraCT Number)
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Participants will receive a single dose of two radio-labelled 6 mg S-770108 capsules (total 12 mg per dose), by oral inhalation using a S-770108 inhaler at a target peak inspiratory flow rate (PIFR) of 15 L/minute on Day 1 of Period 1 followed by a single dose of two radio-labelled 6 mg S-770108 capsules by oral inhalation at a target PIFR of 30 L/minute on Day 1 of Period 2. There will be a 5 to 13 day washout period between the two treatment periods.
  Interventions: Drug: Radio-labelled S-770108; Device: S-770108 Inhaler A1
- Sequence B (Experimental): Participants will receive a single dose of two radio-labelled 6 mg S-770108 capsules (total 12 mg per dose), by oral inhalation using a S- 770108 inhaler at a target PIFR of 30 L/minute on Day 1 of Period 1 followed by a single dose of two radio-labelled 6 mg S-770108 capsules by oral inhalation at a target PIFR of 15 L/minute on Day 1 of Period 2. There will be a 5 to 13 day washout period between the two treatment periods.
  Interventions: Drug: Radio-labelled S-770108; Device: S-770108 Inhaler A1

INTERVENTIONS:
Drug: Radio-labelled S-770108 — 99mTc radio-labelled S-770108 supplied as a capsule containing 6 mg active pirfenidone for inhalation
Device: S-770108 Inhaler A1 — Dry powder inhaler

SUMMARY:
The primary objective of this study is to assess the total lung deposition of radiolabelled S-770108 inhalation powder formulation after each of two separate single inhaled doses in healthy adult participants at two different target peak inspiratory flow rates (PIFRs)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand this study and comply with all study procedures, are able to be trained and use the device correctly at screening and willing to provide written informed consent before screening.
2. Subjects judged to be healthy by the principal or sub investigator, based on medical history and clinical evaluation.
3. Male and female subjects ≥ 40 to ≤ 80 years of age at the time of informed consent.
4. Subjects whose body mass index (BMI) is ≥ 18.0 and < 30.0 kg/m2 during the screening visit．
5. Subjects able to produce a peak inspiratory flow rate of at least 30.00L/min at screening using the investigational device attached to an electronic flow meter.
6. Subjects who have smoked within 12 months before admission cannot be entered the study.
7. Subjects judged to have normal lung function. Specifically, with percent predicted forced expiratory volume in 1 second (%FEV1) ≥ 80% and forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) ratio ≥70%.
8. Male subjects are eligible to participate if they agree to the following during the treatment period and for at least 3 months (a spermatogenesis cycle) after the last dose of study intervention.

   * Refrain from donating sperm.
   * Must agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as described in Appendix 2, as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
9. Female subjects who agree to use of appropriate contraception measures from time of screening until 3 months after the last dose of study drug, except for female subjects who are surgically sterile by bilateral oophorectomy for at least 6 weeks with appropriate documentation or who are post-menopausal (defined as at least 6 months of spontaneous amenorrhea in woman > 45 years with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL at screening, or at least 12 months of spontaneous amenorrhea in woman > 45 years)

Exclusion Criteria:

1. Subjects deemed by the principal or sub investigator to be ineligible for the study due to history of, or concurrent and clinically significant metabolic or endocrine, hepatic, renal, haematological, respiratory, cardiovascular, gastrointestinal, urological, immunological, neurological or psychiatric disorders, or any malignant neoplasms at any diagnosed stage.
2. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2018, shall participate in the study.
3. Subjects who have a history of clinically relevant respiratory disease, diseases affecting respiratory function, E.N.T. diseases, or lung surgery.
4. Subjects who have had an upper respiratory infection in the last 7 days which could affect inhalation/absorption of study medication.
5. Subjects who use regular medication (prescribed and/or over the counter) or have used any medication (excluding non-prescription drugs, vitamins, and dietary or herbal supplements which do not interfere with respiratory function according to their labelling) within 14 days before admission; exceptions may be permitted on a case by case basis if considered not to interfere with the aims of the study and agreed by the investigator and sponsor's medical monitor.
6. Subjects with a history of lactose intolerance, intolerance to dairy products, or a history of gluten intolerance.
7. Subjects with a history of serious adverse reaction or serious hypersensitivity to the active ingredient or excipients in any drug.
8. Subjects with a history of drug and/or alcohol addiction within the past 2 years before screening or a positive test for drugs or alcohol at screening or admission visit.
9. Regular alcohol consumption in males of > 21 units per week, or females of > 14 units per week (1 unit = 1/2 pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
10. Subjects with a positive result on any of the tests for the serologic detection of human immunodeficiency virus (HIV) antigen/antibody, hepatitis B surface antigen (HBsAg), and hepatitis C antibody.
11. Female subjects who are pregnant, breast-feeding, have a positive pregnancy test result during the screening assessment or admissions; or intending to become pregnant during the study period or within 3 months after the last dose of study treatment.
12. Subjects who have donated > 400 mL of blood within 3 months before screening, > 200 mL within 4 weeks before screening, or who donated blood between screening and admission.
13. Subjects who have been exposed to an investigational drug within 90 days prior to study drug administration.
14. Subjects who have previously received pirfenidone (Esbriet®, Pirespa®) in any form, or S 770108.
15. Subjects who are study site employees or immediate family members of a study site employee, or sponsor employees.
16. Subjects who are ineligible for the study for any other reason, as judged by the investigator or sub investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Total lung deposition of 99mTc radio-labelled S-770108 | Day 1 of each treatment period
  Deposition of 99mTc radio-labelled S-770108 in both lungs will be assessed using gamma scintigraphy imaging.

SECONDARY OUTCOMES:
Central lung deposition of 99mTc radio-labelled S-770108 | Day 1 of each treatment period
  Deposition of 99mTc radio-labelled S-770108 in both lungs will be assessed using gamma scintigraphy imaging.
Peripheral lung deposition of 99mTc radio-labelled S-770108 | Day 1 of each treatment period
  Deposition of 99mTc radio-labelled S-770108 in both lungs will be assessed using gamma scintigraphy imaging.
Penetration index of 99mTc radio-labelled S-770108 | Day 1 of each treatment period
  Ratio of peripheral to central deposition, assessed using gamma scintigraphy imaging.
Extra-pulmonary deposition of 99mTc radio-labelled S-770108 | Day 1 of each treatment period
  Extra-pulmonary deposition including stomach deposition, oropharyngeal deposition, retention in the device and capsules, and exhaled air filter deposition.
Number of device deficiencies | Day 1 of each treatment period
  Device Deficiencies are defined as inadequacies of the investigational medical device with respect to its identity, quality, durability, reliability, safety or performance; for example: malfunctions, use errors, and inadequate labelling in the information supplied by the manufacturer.
Number of participants with adverse events | From first dose of study drug to 14 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Simbec-Orion, Merthyr Tydfil, Merthyr Tydfil, United Kingdom